CLINICAL TRIAL: NCT07176650
Title: A Randomized, Multicenter, Double-Blind, Parallel-Controlled, Phase I Clinical Study To Evaluate Pharmacokinetic Profile, Safety, Efficacy and Immunogenicity Of Ipilimumab Biosimilar HLX13 Vs. YERVOY® (US-Sourced YERVOY®) As A First-Line Treatment For Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Phase I Clinical Study To Evaluate Pharmacokinetic Profile, Safety, Efficacy and Immunogenicity Of Ipilimumab Biosimilar HLX13 Vs. YERVOY® (US-Sourced YERVOY®) As A First-Line Treatment For Patients With Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX13-HCC102
Record Dates: First submitted 2025-09-01; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HLX13 Group (Experimental)
  Interventions: Drug: HLX13; Drug: OPDIVO
- US-sourced YERVOY® Group (Active Comparator)
  Interventions: Drug: Yervoy; Drug: OPDIVO

INTERVENTIONS:
Drug: HLX13 — Patients will receive HLX13 (3 mg/kg) treatment on the first day of each 3-week cycle, up to 4 cycles.
  Arms: HLX13 Group
Drug: Yervoy — Patients will receive US-sourced YERVOY® (3 mg/kg) treatment on the first day of each 3-week cycle, up to 4 cycles.
  Arms: US-sourced YERVOY® Group
Drug: OPDIVO — Patients will receive EU-sourced OPDIVO® (EU-sourced nivolumab) (1 mg/kg) treatment on the first day of each 3-week cycle, up to 4 cycles. Subjects who may continue to benefit from OPDIVO® treatment as assessed by investigators will be subsequently treated with local-sourced OPDIVO® monotherapy every 4 weeks, up to 2 year after randomization.

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-controlled, phase I clinical study to evaluate the PK characteristics, safety, efficacy, and immunogenicity of HLX13 and US-sourced YERVOY® in patients with unresectable hepatocellular carcinoma who have not received prior systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed and dated an IRB/IEC-approved written informed consent form (ICF) in accordance with regulatory and institutional guidelines.
2. Male or female, 18 years ≤ age ≤ 65 years at the time of signing the ICF.
3. Body weight: 50 kg-85 kg.
4. Histologically diagnosed hepatocellular carcinoma (HCC); and must have an advanced HCC, defined as: a) not eligible for curative surgical and/or locoregional therapies; or b) progressive disease after surgical and/or locoregional therapies. Subjects with only a radiologic diagnosis of hepatocellular carcinoma may be enrolled for screening in the study but histological confirmation is mandatory prior to randomization.
5. At least one measurable lesion as assessed by investigator based on RECIST v1.1 within 4 weeks prior to the first dose in this study. The measurable lesion is not from sites that have been previously treated with surgery, radiotherapy, and/or locoregional therapy.
6. No systemic therapy for relapsed metastatic or advanced hepatocellular carcinoma prior to screening. Note: prior neo-adjuvant or adjuvant systemic therapy is permitted if recurrence occurs ≥12 months after treatment completion.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 within 7 days prior to the first dose.
8. Cirrhotic status of Child-Pugh Class A within 7 days prior to the first dose.
9. Left ventricular ejection fraction (LVEF) ≥ 50% as measured by echocardiography.
10. Normal major organ functions prior to the first dose.
11. For patients with active hepatitis B virus (HBV), the HBV-DNA must be less than 500 IU/mL or 2500 copies/mL within 28 days prior to the randomization, an anti-HBV treatment (e.g., entecavir) has been started prior to the randomization, and patients are willing to continue the treatment during this study. Patients with positive HCV-RNA must agree to receive standard anti-viral therapy per the local standard of care.
12. Women of childbearing potential should have a negative serum pregnancy test at screening and a negative urine pregnancy test prior to the first dose.

Exclusion Criteria:

1. With other histopathological types of hepatocellular carcinoma, including fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, or mixed cholangiocarcinoma and hepatocellular carcinoma.
2. Other malignancies active within 3 years prior to or at screening except for localized tumors that have been cured such as basal cell carcinoma, squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
3. Liver transplant, or organ allograft or allogeneic bone marrow transplantation prior to screening, or the above transplantation is scheduled during the study.
4. History of hepatic encephalopathy prior to screening.
5. Clinically significant ascites.
6. Patients with tumor thrombus at the main portal vein (Vp4), or inferior vena cava prior to screening, or clear invasion into the bile duct, or HCC with ≥50% liver occupation.
7. Presence of nervous system disorders at screening.
8. Evidence of portal hypertension with bleeding esophageal or gastric varices within 6 months prior to the randomization. The aforementioned patients have undergone endoscopy to exclude those with high hemorrhage risk may be enrolled. For a patient receiving endoscopy within 6 months prior to randomization, repeat examination is not required.
9. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 3 months prior to screening except for esophageal or gastric varices.
10. History of non-healing wounds, bone fractures, or ulcers at risk of bleeding within 3 months prior to randomization.
11. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the randomization or those who receive minor surgical procedures (e.g., core biopsy) within 7 days prior to randomization.
12. Known active or suspected autoimmune diseases prior to screening. Patients with stable disease who do not require systemic immunosuppressive therapy may also participate.
13. Treatment with systemic corticosteroids (> equivalent dose of 10 mg/day prednisone) or other immunosuppressive agents within 14 days prior to the first dose or during the study. However, for patients with conditions other than active autoimmune diseases, inhaled or topical steroids or adrenocortical hormone replacement therapy (no more than the equivalent dose of 10 mg/day prednisone) are allowed.
14. Active co-infection with both hepatitis B and C (or detectable HBV surface antigen or HBV-DNA and HCV-RNA at screening), or hepatitis D infection in subjects with hepatitis B.
15. Subjects with a history of co-infection with both hepatitis B and C.
16. Human immunodeficiency virus (HIV) infection prior to screening (or positive anti-HIV at screening).
17. Any active infections (including, but not limited to bacteria, fungi, mycoplasma, chlamydia, and herpes zoster virus) requiring systemic treatment within 14 days prior to screening.
18. Uncontrolled cardiovascular diseases within 6 months prior to screening.
19. Known interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, and severe lung function abnormalities that may impede the investigators' diagnosis and management of drug-related pulmonary toxicity prior to screening.
20. Patients who have used traditional Chinese herbs or medicines with anti-tumor indications within 14 days prior to randomization.
21. Patients who have received treatment with live vaccines within 28 days prior to randomization. Those who received inactivated viral vaccines for seasonal influenza or COVID-19 are eligible.
22. Patients who have received any T-cell costimulatory agents or immune checkpoint blockade therapy, including but not limited to cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, or other agents that target T cells.
23. Radical radiotherapy within 4 weeks prior to randomization.
24. Other prior/concomitant therapy: a) Treatment with strong CYP3A4 inducers within 1 week prior to randomization, including rifampin (and its analogues) or St. John's wort. b) Use of anticoagulants such as, warfarin or similar agents requiring therapeutic INR monitoring. Note: Treatment with low molecular weight heparin is allowed. c) Treatment with anti platelet therapy (aspirin at dose ≥ 300 mg/day, clopidogrel at dose ≥75 mg/day).
25. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or IMP administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
26. Anaphylaxis to ipilimumab, nivolumab, or any other monoclonal antibody, or any component of the IMPs prior to screening.
27. History of psychotropic substance abuse or illicit drug use as judged by the investigator prior to screening.
28. Pregnant and lactating women, and those intending to become pregnant during the study or within 5 months after the last study treatment.
29. Currently participating in another clinical study prior to screening, or less than 4 weeks or 5 half-lives of the IMPs in the previous study, whichever is longer, between the screening of the study and the end of treatment in the previous study.
30. Patients who have other conditions not suitable for inclusion per investigator's judgments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time 0 to 21 days (AUC0-21d) after the 1st dose | from time 0 to 21 days after the 1st dose (3 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Area under the serum concentration-time curve within a dosing interval at steady-state (AUCss) after the 4th dose | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Maximum serum drug concentration (Cmax) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Maximum serum drug concentration at steady-state (Cmax,ss) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Trough serum drug concentration (Ctrough) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Trough serum drug concentration at steady-state (Ctrough,ss) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum serum drug concentration (Tmax) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to reach maximum serum drug concentration at steady-state (Tmax,ss) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Adverse events (AEs) | From enrollment to the end of 90-day safety follow-up (21 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Serious adverse events (SAEs) | From enrollment to the end of 90-day safety follow-up (21 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Adverse events of special interest (AESIs) | From enrollment to the end of 90-day safety follow-up (21 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal vital signs | From enrollment to the end of 30-day safety follow-up (13 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal physical examination findings | From enrollment to the end of 30-day safety follow-up (13 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal Laboratory tests results (hematology, serum chemistry, endocrine function, coagulation function, and myocardial enzymes) | From enrollment to the end of 30-day safety follow-up (13 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Number of participants with abnormal 12-lead ECG readings | From enrollment to the end of 30-day safety follow-up (13 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Objective response rate (ORR) | From enrollment to the end of treatment (12 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Time to response (TTR) | From enrollment to the end of treatment (12 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Incidence of anti-drug antibody (ADA) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Incidence of neutralizing antibody (NAb) | from time 0 to 78 days after the 4th dose (20 weeks)
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan